CLINICAL TRIAL: NCT05185310
Title: Strategies in Patients Undergoing Repeat AF Ablation
Acronym: TRAP-AF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB # 850051
Record Dates: First submitted 2021-12-20; First posted 2022-01-11 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Atrial Fibrillation
Keywords: pulmonary vein ablation; repeat ablation; posterior wall isolation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: single blinded randomized trial comparing 3 ablation strategies
Who Masked: Participant
Masking Description: patients will be blinded to strategy used
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CTI/AAD (control) (Experimental): In all arms, patients are undergoing first redo AF ablation and the pulmonary veins are chronically isolated and no non-PV triggers elicited during provocation. Arm 1- Cavo-tricuspid isthmus (CTI) ablation with adjustment and/or optimization of antiarrhythmic drug regimen where possible (control arm)
  Interventions: Procedure: Ablation
- Posterior wall isolation (Experimental): In all arms, patients are undergoing first redo AF ablation and the pulmonary veins are chronically isolated and no non-PV triggers elicited during provocation. Arm 2-LA Posterior wall isolation by creation of a LA roof and floor line
  Interventions: Procedure: Ablation
- Empiric Isolation of common trigger sites (Experimental): In all arms, patients are undergoing first redo AF ablation and the pulmonary veins are chronically isolated and no non-PV triggers elicited during provocation. Arm 3-empiric ablation of common sites of non-PV triggers of AF in both the right and left atria.
  Interventions: Procedure: Ablation

INTERVENTIONS:
Procedure: Ablation — Ablation strategy during repeat AF ablation

SUMMARY:
The aim of the proposed research project is to compare the efficacy of three different ablation strategies in patients with atrial fibrillation (AF) who are undergoing their first repeat catheter ablation for recurrent AF.

DETAILED DESCRIPTION:
Reconnection of the pulmonary veins (PV) is generally responsible for AF recurrence in most cases. However, in a growing subset of patients undergoing repeat ablation for recurrent AF, the PVs are chronically isolated and no other non-PV triggers of AF can be identified. The investigators have previously shown that empirically ablating at known common non-PV trigger sites for AF can improve arrhythmia free survival beyond PVI. The left atrial (LA) posterior wall is also increasingly being isolated in AF patients undergoing catheter ablation. However, long term arrhythmia free survival in AF patients undergoing LA posterior wall isolation is not consistently better than PVI alone.

The objective of this study therefore is to assess whether performing empiric ablation of common non-PV trigger sites or achieving LA posterior wall isolation can improve arrhythmia free survival in AF patients who are undergoing repeat AF ablation and in whom the PV remain chronically isolated and/or do not demonstrate AF. The investigators propose to do this as prospective, randomized three arm study.

ELIGIBILITY:
Inclusion Criteria: All patients undergoing first redo AF ablation who have chronically isolated pulmonary veins and no non-PV triggers with provocation testing (randomized intra-procedure).

Exclusion Criteria:

1. Patients in whom ≥1 PVs have reconnected and AF triggers can be elicited from the reconnected PV.
2. Patients who demonstrated non-PV triggers for AF.
3. Patients who have experienced arrhythmia recurrence post ablation where the recurrent arrhythmia is other than atrial fibrillation or typical atrial flutter
4. Failure to obtain informed consent
5. Patients with a mechanical mitral valve

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-12-13 (Actual); Primary Completion 2023-02-03 (Actual); Study Completion 2023-02-03 (Actual)

PRIMARY OUTCOMES:
Primary efficacy endpoint | 1 year
  Freedom from atrial arrhythmias off antiarrhythmic medications at 1 year after 1 repeat ablation procedure. Subjects are seen at 6 weeks, 6 months and 1 year post procedure with ECG at each visit and monitors at 6 months and one year to assess efficacy. Information regarding medications, health status, arrhythmia symptoms, and ECG and monitor results documented.

SECONDARY OUTCOMES:
Secondary endpoint | 1 year
  Composite: Freedom from atrial arrhythmias at 1 year after 1 repeat ablation procedure off antiarrhythmic medications; AF related interventions and hospitalizations (electrical cardioversion, increase or change in antiarrhythmic medication, repeat ablation, hospitalization for complication, etc). Subjects are seen at 6 weeks, 6 months and 1 year post procedure with ECG at each visit and monitors at 6 months and one year to assess efficacy. Information regarding medications, health status, hospitalizations (including repeat ablations and cardioversion), arrhythmia symptoms, and ECG and monitor results documented.

CONTACTS AND LOCATIONS:
Overall Officials: David Lin, MD, Principal Investigator — University of Pennsylvania; Sanjay Dixit, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided